CLINICAL TRIAL: NCT04975984
Title: Evaluation of Expectant Management in Women Diagnosed With a Tubal Ectopic Pregnancy at Ain-Shams University Maternity Hospital Over the Period From January 1, 2016 to December 31, 2020
Brief Title: Expectant Management of Ectopic Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, associate professor, Ain Shams University
Other Study IDs: ASU FM1
Record Dates: First submitted 2021-06-17; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: qualitative hCG levels and ultrasound criteria — detect upper limit of qualitative hCG levels associated with successful expectant management of ectopic pregnancy

SUMMARY:
The aim of this study is to assess the efficacy and safety of expectant management in the treatment of tubal ectopic pregnancy and identification of different factors that can be used to predict its success.

ELIGIBILITY:
Inclusion Criteria:

- all women who underwent expectant management as the first line of management offered after optimal counseling during the period from January 1, 2016 to December 31, 2020.

1. Hemodynamically stable with confirmed diagnosis of ectopic pregnancy on ultrasound scan.
2. No significant pelvic pain.
3. No hemoperitoneum.
4. No fetal heart in the ectopic pregnancy.
5. HCG level <5000 IU/L.
6. Expectant management was the first line of management offered to the patient after optimal counseling.

Exclusion Criteria:

1. all women with non tubal ectopic pregnancy
2. all women with tubal ectopic pregnancy that recieved medical or surgical treatment as 1st line treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants included in this study will have the following criteria:
  1. Hemodynamically stable with confirmed diagnosis of ectopic pregnancy on ultrasound scan.
  2. No significant pelvic pain.
  3. No hemoperitoneum.
  4. No fetal heart in the ectopic pregnancy.
  5. HCG level <5000 IU/L.
  6. Expectant management was the first line of management offered to the patient after optimal counseling.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-20 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
resolution of hCG level | up to 12 weeks
  hCG levels measured every week till negative less than (<20 IU/l) up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No